CLINICAL TRIAL: NCT06684717
Title: Using an Educational Video to Enhance Adherence of Continuous Positive Pressure Therapy in Thai Obstructive Sleep Apnea Patients: a Randomised Controlled Trial
Brief Title: Using an Educational Video to Enhance Adherence of CPAP Therapy in Thai OSA Patients: a Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Jindapa Srikajon, MD., Siriraj Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 042/2566(IRB2)
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: OSA

STUDY DESIGN:
Intervention Model Description: Inclusion criteria were adults (older than age 18) who were diagnosed with moderate to severe OSA or mild OSA with an indication for CPAP therapy by standard polysomnography (PSG) from 1 December 2022 and 31 May 2023 at Siriraj sleep center. Diagnosis of obstructive sleep apnea (OSA) was done according to the AASM criteria; mild (AHI 5 to ≤ 15 events/h), moderate (AHI 15 to ≤ 30 events/h) and severe (AHI ≥ 30 events/h). Subjects who were not CPAP naïve had central sleep apnea, had comorbidities that were contraindicated for CPAP therapy, or denied using CPAP were excluded.
Who Masked: Investigator
Masking Description: Random permuted blocks design was used to randomly assign each participant into video education intervention and usual care group by a research assistant, without the principal investigator knowing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational video intervention group (Experimental): The participants who were randomized into the video group watched a 3-minute video that educated patients about OSA, treatment, and its benefits. We also added the scenario of the real patients who were currently using CPAP, in order to motivated participants to use CPAP more. The participants in the video group also received routine care.
  Interventions: Behavioral: Educational video intervention
- Usual care group (No Intervention): In the usual care group, they were routinely advised about the disease and CPAP machine use by sleep medicine doctors and sleep technicians.

INTERVENTIONS:
Behavioral: Educational video intervention — A 3-minute educational video mainly about the benefits of Continuous positive airway pressure therapy in OSA patients. The video starts with basic knowledge about OSA and how it affects human health. What is a CPAP machine and how does it works? It was developed from consensus among expert opinions of Neurobehavioral specialists and sleep physicians.
  Arms: Educational video intervention group

SUMMARY:
The goal of this clinical trial is to find out whether video education helps improve CPAP adherence in OSA patients or not

The main questions it aims to answer are:

Does educational video intervention help improve CPAP adherence in Thai OSA patients? What factors predict good CPAP adherence in OSA patients?

Participants will:

be randomized into video intervention group and usual care group with simple random sampling method. Demographics, Epworth Sleepiness scale scores (ESS), Pittsburg sleep quality scores, polysomnographic data and CPAP usage data were recorded.

DETAILED DESCRIPTION:
INTRODUCTION

The prevalence of obstructive sleep apnea (OSA) is increasing globally. Continuous positive airway pressure (CPAP) therapy is the most frequently used and effective treatment for moderate and severe OSA. It has been proven to improve sleep quality and decrease cardiovascular events, such as stroke and myocardial infarction.

When treating OSA with CPAP, one essential obstacle is the challenge of obtaining adequate compliance. Good compliance is defined as use during at least 4 h/night and for more than 70% of nights. It appeared that the longer nightly uses is associated with better functional outcomes such as daytime sleepiness. Best results for quality of life improvements and optimal reductions in blood pressure also occur when CPAP usage ≥ 4 h/night. However, the previous data demonstrated subjective adherence ranges of 65%-90%, whereas objective measures of CPAP adherence demonstrated use in the range of 40%-83%. There were various interventions to improve CPAP adherence including education, behavioral, technological, and supportive strategies. Among all, education strategy remains the most consistent intervention in CPAP naïve patients, since the common causes of poor CPAP adherence are patients' negative perceptions of the benefit and health value of CPAP and also lack of confidence in the therapeutic effect of CPAP results. From the previous study, systemic education tends to improve adherence approximately 35 to 50 minutes per night. According to the American Academy of Sleep Medicine Clinical Practice Guideline for Treatment of Adult OSA with Positive Airway Pressure (PAP), strongly recommend that educational interventions be given prior to initiation of PAP therapy in adults with OSA. Wiese et al. found that OSA patients with educational video intervention had a higher rate of return at the clinic. However, objective CPAP adherence was not available most of patients. It is shown that the adherence rate to CPAP therapy tends to be improved by visual education although not significant in a study by Basoglu et al.

In recent study which assessed the impact of a video on CPAP adherence in a population of patients at increased risk for poor CPAP adherence, the results were not significant. Despite the insignificant results of the previous studies, we still decided to evaluate the impact of educational videos on CPAP usage in Thai patients which is low cost and requires lower manpower. To the best of our knowledge, this is the first study about the effectiveness of video education in CPAP adherence improvement in the Thai population.

The primary aim of this study was to find out whether video education would benefit CPAP adherence rate in OSA patients or not.

MATERIALS AND METHODS Participants This was a randomized controlled trial study. Inclusion criteria were adults (older than age 18) who were diagnosed with moderate to severe OSA or mild OSA with indication for CPAP therapy by standard polysomnography (PSG) from 1 December 2022 and 31 May 2023 at Siriraj sleep center. Diagnosis of obstructive sleep apnea (OSA) was done according to the AASM criteria; mild (AHI 5 to ≤ 15 events/h), moderate (AHI 15 to ≤ 30 events/h) and severe (AHI ≥ 30 events/h). Subjects who were not CPAP naïve, had central sleep apnea, had comorbidities which were contraindicated for CPAP therapy or denied using CPAP were excluded. Sample size calculation was done based on previous studies and expert opinion from our research team discussion. An estimated total sample size was 132. Procedure

1. Enrolled patients were informed about the study and asked for consent form on the date of appointment after PSG study. 5
2. The demographic data and PSG study result were recorded. The Epworth Sleepiness Scale (ESS), Fatigue Severity Scale(FSS) and Pittsburg Sleep Quality Index(PSQI) were also obtained.
3. Random permuted blocks design was used to randomly assigned each participant into video education intervention and usual care group.
4. The participants who were randomized into the video group watched a 3 minute video which educated patients about OSA, treatment and its benefits. We also added the scenario of the real patients who were currently using CPAP, in order to motivated participants to use CPAP more. The participants in the video group also received routine usual care.
5. In the usual care group, they were routinely advised about the disease and CPAP machine use by sleep medicine doctors and sleep technicians.
6. After prescribed with CPAP therapy, all patients were appointed to return at 3 weeks.
7. CPAP usage data and sleep questionnaire were collected at 3 weeks. Outcome Analysis The primary outcome was percent meeting previous criteria for good adherence (2) at 3 weeks in video intervention group compared to usual care group. Usage data for the past 3 weeks was retrieved from the device memory card. While the secondary outcome were average CPAP usage all days (hours per night) at 3 weeks in video intervention group compared to usual care group, the % of days with an CPAP usage of ≥4 h at 3 weeks in video intervention group compared to usual care. The study was approved by the Human research ethics committee of Siriraj hospital, Mahidol university (SIRB protocol No. 042/2566).

STATISTICAL ANALYIS Descriptive statistical analysis was performed using the SPSS 20.0. Continuous variables were expressed as mean and standard deviation while categorical variables were expressed as number and percentage. Comparisons between groups were carried out with Mann-Whitney U test or Student's t-test. Categorical variables were compared with the chi-square test. Statistical significance was considered as p-value less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Participants who were diagnosed with moderate to severe OSA or mild OSA with indication for CPAP therapy by standard polysomnography (PSG) from 1 December 2022 and 31 May 2023 at Siriraj Sleep Center. Diagnosis of obstructive sleep apnea (OSA) was done according to the AASM criteria; mild (AHI 5 to ≤ 15 events/h), moderate (AHI 15 to ≤ 30 events/h) and severe (AHI ≥ 30 events/h).

Exclusion Criteria:

* Participants who were not CPAP naïve, had central sleep apnea, had comorbidities that were contraindicated for CPAP therapy or denied using CPAP.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2024-02-17 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
CPAP adherence rate at 3 weeks after intervention. | 3 weeks
  The percent of participants meeting the criteria for good CPAP adherence (more than 4 hours per night and more than 70% of all days used) at 3 weeks in the video intervention group compared to the usual care group. Usage data for the past 3 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No